CLINICAL TRIAL: NCT00658788
Title: A Multi-Center, Open-Label Study to Evaluate the Safety and Efficacy of a Consecutive Treatment Regimen of Clobetasol Propionate 0.05% Spray, Followed by Calcitriol Ointment 3µg/g, in the Management of Moderate to Severe Plaque Psoriasis
Brief Title: Safety & Effectiveness of Clobex Spray, Followed by Calcitriol Ointment in Management of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US10085
Record Dates: First submitted 2008-03-04; First posted 2008-04-15 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2012-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Treatment (Active Comparator): clobetasol propionate spray 0.05%
  Other Names:
  Clobex® Spray 0.05% clobetasol propionate spray, 0.05%, applied topically twice daily
  calcitriol ointment
  Other Names:
  Calcitriol Ointment calcitriol ointment, 3 µg/g, applied topically, not to exceed 30 g daily
  Interventions: Drug: clobetasol propionate spray 0.05%; Drug: calcitriol ointment

INTERVENTIONS:
Drug: clobetasol propionate spray 0.05% — clobetasol propionate spray, 0.05%, applied topically twice daily
  Other Names: Clobex® Spray 0.05%
Drug: calcitriol ointment — calcitriol ointment, 3 µg/g, applied topically, not to exceed 30 g daily

SUMMARY:
The primary objectives of this study are to evaluate the safety & efficacy of consecutive treatments of Clobex® Spray and Silkis® Ointment in the management of plaque psoriasis.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe plaque psoriasis, defined as 3% - 20% treatable body surface area
* Overall Disease Severity of at least 3 (moderate)

Exclusion Criteria:

* Surface area involvement too large (>20% BSA)
* Psoriasis involving only the scalp, groin, axillae, and/or other intertriginous areas

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (12):
- United States (12):
  - Therapeutics Clinical Research, San Diego, California
  - MedaPhase, Inc., Newnan, Georgia
  - Gwinnett Clinical Research Center, Inc, Snellville, Georgia
  - Hudson Dermatology, Evansville, Indiana
  - Mount Sinai Department of Dermatology, New York, New York
  - Northeastern Ohio Universities College of Medicine, Warren, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - J&J Studies, Inc, College Station, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Dermatology Associates of Seattle, PLLC, Seattle, Washington
  - Madison Skin and Research, Inc, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequential Treatment Regimen: 4 weeks Clobex® Spray 0.05% Treatment Applied Topically Twice Daily Followed by Calcitriol Ointment, 3 µg/g Applied Once Daily
Period: Overall Study
Arm/Group | Sequential Treatment Regimen
Started | 305
Completed | 231
Not Completed | 74
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 18
Not completed — Treatment Discontinuation | 32

BASELINE CHARACTERISTICS:
Arm/Group | Sequential Treatment Regimen
Number analyzed (Participants) | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 278
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 273
  More than one race | 12
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Disease Severity Success (ODS)
Description: Success was defined as a one-grade improvement in ODS from baseline.
Time Frame: 8 and 12 weeks
Population: The per protocol population included 170 subjects who completed the 12 week regimen without any major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sequential Treatment Regimen
Number analyzed (Participants) | 170
percentage of participants
  Week 8 | 100.0 [97.9 to 100.0]
  Week 12 | 84.1 [77.7 to 89.3]

2. Secondary Outcome: Global Improvement Score
Time Frame: 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Groups:
- Week 2; Week 4; Week 8; Week 12: 4 weeks Clobex® Spray 0.05% Treatment Applied Topically Twice Daily Followed by 8 Weeks of Calcitriol Ointment, 3 µg/g Applied Once Daily
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 170 | 170 | 170 | 170
participants
  -1:Symptoms | 1 | 0 | 0 | 0
  0:No Change | 4 | 2 | 10 | 13
  1:Minimal Improvement | 9 | 4 | 12 | 19
  2:Definite Improvement | 53 | 26 | 43 | 49
  3:Considerable Improvement | 93 | 96 | 77 | 58
  4:Clearing | 11 | 42 | 28 | 31

3. Secondary Outcome: Signs of Psoriasis - Erythema
Time Frame: 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 170 | 170 | 170 | 170
participants
  Clear | 0 | 9 | 13 | 12
  Almost Clear | 46 | 81 | 53 | 41
  Mild | 82 | 57 | 70 | 60
  Moderate | 35 | 23 | 32 | 53
  Severe/Very Severe | 7 | 0 | 2 | 4

4. Secondary Outcome: Signs of Psoriasis - Scaling
Time Frame: 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 170 | 170 | 170 | 170
participants
  Clear | 25 | 41 | 36 | 31
  Almost Clear | 61 | 83 | 53 | 56
  Mild | 63 | 37 | 71 | 54
  Moderate | 19 | 9 | 9 | 26
  Severe/Very Severe | 4 | 0 | 1 | 3

5. Secondary Outcome: Signs of Psoriasis - Plaque Elevation
Time Frame: 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 170 | 170 | 170 | 170
participants
  Clear | 22 | 46 | 35 | 24
  Almost Clear | 69 | 78 | 50 | 45
  Mild | 54 | 36 | 68 | 61
  Moderate | 24 | 9 | 17 | 39
  Severe/Very Severe | 1 | 1 | 0 | 1

6. Secondary Outcome: Percent Change From Baseline in Body Surface Area (% BSA) Affected
Time Frame: 2, 4, 8 and 12 weeks
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 170 | 170 | 170 | 170
Percent Change from Baseline | 20.1 (23.6) | 43.1 (30.9) | 46.6 (31.1) | 46.2 (36.1)

7. Secondary Outcome: Overall Disease Severity
Time Frame: 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 170 | 170 | 170 | 170
participants
  Clear | 0 | 5 | 9 | 11
  Almost Clear | 53 | 100 | 60 | 45
  Mild | 83 | 53 | 88 | 70
  Moderate | 31 | 12 | 13 | 44
  Severe/Very Severe | 3 | 0 | 0 | 0

8. Secondary Outcome: Tolerability Assessment - Pruritus
Time Frame: Baseline, 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Groups:
- Baseline; Week 2; Week 4; Week 8; Week 12: 4 weeks Clobex® Spray 0.05% Treatment Applied Topically Twice Daily Followed by 8 Weeks of Calcitriol Ointment, 3 µg/g Applied Once Daily
Arm/Group | Baseline | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 305 | 288 | 285 | 274 | 235
participants
  None | 74 | 179 | 220 | 172 | 128
  Mild | 84 | 91 | 56 | 66 | 65
  Moderate | 84 | 13 | 9 | 31 | 32
  Severe | 63 | 5 | 0 | 5 | 10

9. Secondary Outcome: Tolerability Assessment - Telangiectasias
Time Frame: Baseline, 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 305 | 288 | 285 | 274 | 235
participants
  None | 303 | 284 | 283 | 273 | 230
  Mild | 1 | 4 | 2 | 1 | 5
  Moderate | 0 | 0 | 0 | 0 | 0
  Severe | 1 | 0 | 0 | 0 | 0

10. Secondary Outcome: Tolerability Assessment - Stinging/ Burning
Time Frame: Baseline, 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 305 | 288 | 285 | 274 | 235
participants
  None | 200 | 232 | 245 | 234 | 200
  Mild | 44 | 42 | 34 | 18 | 24
  Moderate | 31 | 13 | 4 | 19 | 8
  Severe | 30 | 1 | 1 | 3 | 3

11. Secondary Outcome: Tolerability Assessment - Skin Atrophy
Time Frame: Baseline, 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 305 | 288 | 285 | 274 | 235
participants
  Absent | 303 | 286 | 278 | 270 | 233
  Present | 2 | 2 | 7 | 4 | 2

12. Secondary Outcome: Tolerability Assessment - Folliculitis
Time Frame: Baseline, 2, 4, 8 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 305 | 288 | 285 | 274 | 235
participants
  Absent | 303 | 286 | 274 | 271 | 232
  Present | 2 | 2 | 11 | 3 | 3

ADVERSE EVENTS:
Arm/Group | Sequential Treatment Regimen
Serious Adverse Events (participants affected / at risk) | 9/305
Other Adverse Events (participants affected / at risk) | 0/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sequential Treatment Regimen (N=305)
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Hemiplegia (Nervous system disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days